CLINICAL TRIAL: NCT03217955
Title: Cognitive Behavioural Therapy- Social Functioning In Adolescence With Recent Onset Schizophrenia
Acronym: Social
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Arkin (Industry); Vroege Psychose ABC - Utrecht (Unknown); Centrum Eerste Psychose, Utrecht, Netherlands (Unknown); GGZ inGeest (Other)
Responsible Party: Principal Investigator, Lieuwe de Haan, PhD, Professor of Psychotic Disorders, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL46776.018.13
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The present study entails a single-blind two-level RCT directed at patients with recent onset schizophrenia. Participants are randomly assigned to intervention condition (Cognitive Behavioral Therapy- Social Activation (CBTsa) plus Standard Treatment (ST)), or to the control condition (ST alone).
  A baseline test battery is employed to examine causes of social withdrawal and interaction with treatment outcome. Follow-up assessments (repetition test battery) will take place directly after the intervention period and 6 months post-treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomisation is coordinated a staff member of the psychosis department who is not involved in the research team and not familiar with both the assessments or intervention procedure. The results of the randomization is concealed from the assessors. Every effort has been made to keep assessors blind to treatment condition, using the following strategies: research workers were not involved in the randomization process, therapists and research workers made use of different (secured) agendas, and work locations / rooms in order tot minimize the chance of potential blind breaks; patients will be frequently reminded by assessors not to talk about treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-SA (Experimental): 1. Group sessions for 4 weeks, two sessions per week, 60 minutes per session, two trainers (a CBT therapist and a CBT assistant); eight participants, and;
  2. Individual sessions (crystallizing learned skills, focus on individual needs) during 6-8 weeks, one session per week, 45 minutes per session
  Interventions: Behavioral: CBT-SA; Behavioral: Standard Treatment
- Standard Treatment (Active Comparator): Participants in both study conditions will receive ST. Participants are hospitalized or attending day-treatment at the Department of Early Psychosis, Amsterdam, the psychosis department of the ABC team, Utrecht, Parnassia Den Haag and collaborating (local community) mental health centers.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: CBT-SA — Info has been included in arm description
  Arms: CBT-SA
Behavioral: Standard Treatment — Info has been included in arm description

SUMMARY:
Rationale: There is growing consensus that targeting negative symptoms such as social withdrawal is essential to be able to preserve social participation, thereby reducing the high yearly costs of schizophrenia. Aaron T. Beck, founder of Cognitive Behavioural Therapy (CBT), and colleagues have developed and investigated a new CBT approach, in which they target inactivity in a chronic schizophrenia population with severe negative symptoms The therapy is based on accumulating evidence that dysfunctional beliefs in conjunction with neurocognitive impairments can impede social functioning. These results suggest that CBT can be highly successful in establishing clinically meaningful improvements. However, the therapy has not yet been investigated in a recent-onset population.

Objective: To evaluate the applicability and (cost-) effectiveness of a shortened, partly group based, Cognitive Behavioural Therapy focussing on social activation (CBTsa) in patients with recent onset schizophrenia.

Hypotheses: 1) the investigators hypothesized that CBT focused on social activation (CBTsa) in a recent-onset population will result in a substantial reduction in severity of negative symptoms, in particular social withdrawal.

2) The investigators expected that CBTsa would lead to an improvement in terms of Quality of Life and overall functioning.

3) The investigators expected this intervention to result in a reduction in need for care and QALY gain as a consequence of improvement in symptoms and social functioning.

Study design: Single blind randomized controlled trial with 6 month-follow up. Study population: Patients between 18 and 35 years old with negative symptoms of at least moderate severity, and who have been recently (< 2yrs) diagnosed with schizophrenia.

Intervention (if applicable): Individual and group-based CBT intervention targeting social withdrawal.

Main study parameters/endpoints: Change in negative symptoms, Social functioning, and quality of life, Productivity losses.

DETAILED DESCRIPTION:
There is growing consensus that targeting negative symptoms such as social withdrawal is essential to be able to preserve social participation; thereby reducing the high yearly costs of schizophrenia.

Aaron T. Beck, founder of Cognitive Behavioural Therapy (CBT), and colleagues have developed and investigated a new CBT approach, in which they target inactivity in a chronic schizophrenia population with severe negative symptoms; a subgroup that has always believed to be highly treatment resistant. The therapy is based on accumulating evidence that dysfunctional beliefs in conjunction with neurocognitive impairments can impede functioning. Its primary focus is to help patients overcome isolation and inactivity, thereby improve quality of life, rather than primarily focussing on the reduction of psychotic symptoms. Grant, Beck and colleagues found that patients treated with CBT not only showed more improvement in global functioning than patients in the Standard Treatment condition, they also showed a greater reduction in avolition/apathy and psychotic symptoms. These results suggest that CBT can be highly successful in establishing clinically meaningful improvements.

Thus far, this intervention had only been investigated in patients with chronic schizophrenia although there is increasing evidence that social withdrawal is also prominent in the early phase of the illness. Moreover, there is growing consensus that early intervention is more effective in improving illness course than intervention at a later stage of the illness.

In the present study the investigators aimed to examine whether a relatively short, partly group based CBT targeting negative symptoms in recent-onset schizophrenia patients results in reduced social withdrawal, need for care and improvement in quality of life and in overall functioning compared to treatment as usual.

Primary Objective:

The primary aim of this project was to examine a shortened (+/- 20 sessions) and partly group-based version of the new and promising CBT approach tested in a chronic population (from now: 'Cognitive Behavioural Therapy - Social Activation' (CBTsa)), for its applicability and effectiveness in a recent-onset population. The CBTsa has been adjusted to the specific needs of the young recent-onset cohort.

Secondary Objective(s):

A secondary aim was explore the cost-effectiveness of this new intervention (i.e. the balance between costs and health outcomes for CBTsa compared with treatment as usual(ST).

Hypotheses:

1. CBT focused on social activation (CBTsa) will result in a substantial reduction in severity of negative symptoms, and in particular social withdrawal
2. The intervention will result in a reduction in need for care and QALY gain as a consequence of improvement in symptoms and social functioning.
3. CBTsa will lead to an improvement in terms of Quality of Life and overall functioning and symptomatology.

Study Design The present study entails a single-blind two-level RCT directed at patients with recent onset schizophrenia. Participants will be randomly assigned to intervention condition (Cognitive Behavioral Therapy- Social Activation (CBTsa) plus Standard Treatment (ST)), or to the control condition (ST alone). Patients will be stratified by sex, as females with recent onset schizophrenia have a better prognosis and may respond differentially to CBTsa. A baseline test battery will be employed to examine causes of social withdrawal and interaction with treatment outcome. Follow-up assessments (repetition test battery) will take place directly after the intervention period and 6 months post-treatment.

Study population/ datasources Study sample: patients hospitalized or attending day-treatment or receiving outpatient care at one of the participating centers. To maximize engagement, group therapy will be incorporated in the day program. Individual therapy sessions will be delivered flexibly (time, location). All participants are embedded within a low-threshold intensive outreaching care system (aligned with our academic department).

ELIGIBILITY:
Inclusion Criteria:

1. recent onset schizophrenia or related disorder (start antipsychotic medication <2 yr);
2. Social withdrawal (> 3 moderate severity on the PANSS N4; Passive/apathic social withdrawal; range 0-7);
3. Aged 18-35 years;
4. Fluent in Dutch
5. IQ>70;
6. Able and willing to give informed consent

Exclusion Criteria:

1. Younger than eighteen years of age;
2. No mastery of the Dutch language;
3. Negative symptoms as a consequence of positive symptoms (e.g. withdrawal due to paranoid delusions). Positive symptoms as such are not an exclusion criterion; only when they are considered to be the primary cause of the negative symptoms, in which case CBT focused on positive symptoms or another type of intervention for positive symptoms is called for.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Level of social engagement | 3 months (at study completion)
  Level of social engagement as measured by experiences sampling method
Negative symptoms | 3 months (at study completion)
  Negative symptoms as measured with PANSS
Negative symptoms | 3 months (at study completion)
  Negative symptoms as measured with BNSS

SECONDARY OUTCOMES:
Quality of Life | 3 months (at study completion)
  Assessed with the AQoL
Global functioning | 3 months (at study completion)
  Assessed with the GAF
Productivity losses | 3 months (at study completion)
  Effects on ability to perform paid and unpaid work
Positive and General Symptomatology | 3 months (at study completion)
  As assessed with the PANSS
Depression | 3 months (at study completion)
  Depression as assessed with the Calgary Depression Scale for Schizophrenia
Inhibition/ Activation | 3 months (at study completion)
  Behavioural Inhibition/ Behavioural Activation Scales (BISBAS)
Need for care | 3 months (at study completion)
  Camberwell Assessment of Need

CONTACTS AND LOCATIONS:
Overall Officials: Lieuwe de Haan, Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

REFERENCES:
- [Background] Staring AB, Ter Huurne MA, van der Gaag M. Cognitive Behavioral Therapy for negative symptoms (CBT-n) in psychotic disorders: a pilot study. J Behav Ther Exp Psychiatry. 2013 Sep;44(3):300-6. doi: 10.1016/j.jbtep.2013.01.004. Epub 2013 Feb 1. PMID 23454550
- [Background] Grant PM, Huh GA, Perivoliotis D, Stolar NM, Beck AT. Randomized trial to evaluate the efficacy of cognitive therapy for low-functioning patients with schizophrenia. Arch Gen Psychiatry. 2012 Feb;69(2):121-7. doi: 10.1001/archgenpsychiatry.2011.129. Epub 2011 Oct 3. PMID 21969420
- [Background] Verma S, Subramaniam M, Abdin E, Poon LY, Chong SA. Symptomatic and functional remission in patients with first-episode psychosis. Acta Psychiatr Scand. 2012 Oct;126(4):282-9. doi: 10.1111/j.1600-0447.2012.01883.x. Epub 2012 May 23. PMID 22616617
- [Derived] Wijnen BFM, Pos K, Velthorst E, Schirmbeck F, Chan HY, de Haan L, van der Gaag M, Evers SMAA, Smit F. Economic evaluation of brief cognitive behavioural therapy for social activation in recent-onset psychosis. PLoS One. 2018 Nov 12;13(11):e0206236. doi: 10.1371/journal.pone.0206236. eCollection 2018. PMID 30419038